CLINICAL TRIAL: NCT01429532
Title: Clinical Evaluation of Three Incision-size-dependent Phacoemulsification Systems
Brief Title: Outcomes of 3 Incision-size-dependent Phacoemulsification Systems
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Collaborators: Ministry of Health, China (Other Government); National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Haotian Lin, Department of cataract, Zhongshan Ophthalmic Center, Sun Yat-sen University
Other Study IDs: CCPMOH2010-China2
Record Dates: First submitted 2011-09-04; First posted 2011-09-07 (Estimated); Results first posted 2014-07-11 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-06

CONDITIONS: Cataract
Keywords: Cataract
MeSH Terms: conditions — Cataract | interventions — Phacoemulsification

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Group I: 1.8-mm-incision-size phacoemulsification system
  Interventions: Procedure: phacoemulsification
- Group II: 2.2-mm-incision-size phacoemulsification system
  Interventions: Procedure: phacoemulsification
- Group III: 3.0-mm-incision-size phacoemulsification system
  Interventions: Procedure: phacoemulsification

INTERVENTIONS:
Procedure: phacoemulsification — Cataract surgery performed with three incision-size-dependent phacoemulsification systems (1.8, 2.2 and 3.0 mm)
  Other Names: Three incision-size(1.8, 2.2 and 3.0 mm)

SUMMARY:
The purpose of this study is to compare the outcomes of cataract surgery performed with three incision-size-dependent phacoemulsification systems (1.8, 2.2 and 3.0 mm).

DETAILED DESCRIPTION:
It is generally the case that smaller corneal cataract surgical incisions are associated with more rapid wound healing, more stable corneal biomechanical properties and less surgically induced astigmatism (SIA). With the development of phacoemulsification and foldable intraocular lenses (IOL) during recent decades, the size of clear corneal incisions has been reduced from 3.2-mm (coaxial small incision) to 1.4-mm (bimanual micro incision). Micro incision cataract surgery (MICS), including bimanual and micro coaxial phacoemulsification, has attracted much interest recently, due to its safety and ease of learning. However, the superiority of coaxial micro incision cataract surgery as compared conventional coaxial cataract surgery is still not certain, because micro incision phacoemulsification may result in longer ultrasound time (UST), the use of more ultrasonic power and consequently higher endothelial cell loss (ECL).

In our previous studies of the OZil Torsional phacoemulsification system (Infinity, Alcon), we reported that the safety and effectiveness of cataract surgery are influenced by many factors, including the blade used to create the incision, the phacoemulsification apparatus, and the IOL and mode of IOL delivery, which together constitute a surgical system, whose outcomes are restricted by the best performance of each component. Today, micro coaxial phacoemulsification is in wide use for cataract surgery, but the lower limits of incision size should be understood in the context of the various components of the surgical system.

In this study, we compared the safety and efficacy of three different incision-size-dependent phacoemulsification systems, 1.8, 2.2 and 3.0 mm, and evaluated the relationship between incision size and SIA.

ELIGIBILITY:
Inclusion Criteria:

* age between 55 and 85 years
* the presence of nuclear or cortex-nuclear cataract, grades 2.0 to 4.0 (Lens Opacities Classification System III)
* a transparent central cornea
* pupil dilating to >= 7 mm at the time of preoperative examination
* a preoperative central endothelial cell count of >= 1500 cells per square millimeter

Exclusion Criteria:

* previous intraocular surgery
* glaucoma
* pseudoexfoliation
* uveitis
* high myopia
* diabetes mellitus

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective randomized study comprised 120 patients (120 eyes) with age-related cataract enrolled for surgeries between July 2010 and January 2011 at the Zhongshan Ophthalmic Center, Guangzhou, China.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2010-07; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yizhi Liu, M.D.,Ph.D., Study Director — Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen U, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Weikert MP. Update on bimanual microincisional cataract surgery. Curr Opin Ophthalmol. 2006 Feb;17(1):62-7. doi: 10.1097/01.icu.0000193069.32369.e1. PMID 16436926
- [Background] Alio JL, Agdeppa MC, Rodriguez-Prats JL, Amparo F, Pinero DP. Factors influencing corneal biomechanical changes after microincision cataract surgery and standard coaxial phacoemulsification. J Cataract Refract Surg. 2010 Jun;36(6):890-7. doi: 10.1016/j.jcrs.2009.12.041. PMID 20494758
- [Background] Elkady B, Pinero D, Alio JL. Corneal incision quality: microincision cataract surgery versus microcoaxial phacoemulsification. J Cataract Refract Surg. 2009 Mar;35(3):466-74. doi: 10.1016/j.jcrs.2008.11.047. PMID 19251139
- [Result] Liu Y, Jiang Y, Wu M, Liu Y, Zhang T. Bimanual microincision phacoemulsification in treating hard cataracts using different power modes. Clin Exp Ophthalmol. 2008 Jul;36(5):426-30. PMID 18939349
- [Result] Liu Y, Zeng M, Liu X, Luo L, Yuan Z, Xia Y, Zeng Y. Torsional mode versus conventional ultrasound mode phacoemulsification: randomized comparative clinical study. J Cataract Refract Surg. 2007 Feb;33(2):287-92. doi: 10.1016/j.jcrs.2006.10.044. PMID 17276271
- [Result] Zeng M, Liu X, Liu Y, Xia Y, Luo L, Yuan Z, Zeng Y, Liu Y. Torsional ultrasound modality for hard nucleus phacoemulsification cataract extraction. Br J Ophthalmol. 2008 Aug;92(8):1092-6. doi: 10.1136/bjo.2007.128504. Epub 2008 Jun 20. PMID 18567650
- [Result] Wang Y, Xia Y, Zeng M, Liu X, Luo L, Chen B, Liu Y, Liu Y. Torsional ultrasound efficiency under different vacuum levels in different degrees of nuclear cataract. J Cataract Refract Surg. 2009 Nov;35(11):1941-5. doi: 10.1016/j.jcrs.2009.05.055. PMID 19878827
- [Result] Xia Y, Liu X, Luo L, Zeng Y, Cai X, Zeng M, Liu Y. Early changes in clear cornea incision after phacoemulsification: an anterior segment optical coherence tomography study. Acta Ophthalmol. 2009 Nov;87(7):764-8. doi: 10.1111/j.1755-3768.2008.01333.x. Epub 2009 Jun 22. PMID 19548882
- [Derived] Luo L, Lin H, He M, Congdon N, Yang Y, Liu Y. Clinical evaluation of three incision size-dependent phacoemulsification systems. Am J Ophthalmol. 2012 May;153(5):831-839.e2. doi: 10.1016/j.ajo.2011.10.034. Epub 2012 Feb 4. PMID 22310081
- See also: Home page of our investigation ophthalmic center — http://www.gzzoc.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This prospective randomized study included 120 patients (120 eyes) with age-related cataract enrolled between July 2010 and January 2011 at the Zhong-shan Ophthalmic Center, Guangzhou, China.
Pre-assignment Details: Potential subjects with previous intraocular surgery, glaucoma, pseudoexfoliation, uveitis, high myopia and diabetes mellitus were excluded from participation in the study.
Period: Overall Study
Arm/Group | Group I | Group II | Group III
Started | 40 | 40 | 40
Completed | 40 | 40 | 40
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group I | Group II | Group III | Total
Number analyzed (Participants) | 40 | 40 | 40 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 12 | 36
  >=65 years | 28 | 28 | 28 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.95 (6.05) | 71.37 (7.19) | 72.48 (6.15) | 72.59 (6.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 22 | 21 | 62
  Male | 21 | 18 | 19 | 58
Region of Enrollment [Number; unit: participants]
  China | 40 | 40 | 40 | 120

OUTCOME MEASURES:

1. Primary Outcome: Central Cornea Endothelial Cell Loss
Description: Central cornea endothelial cell loss was calculated on the basis of preoperative and postoperative endothelial cell density.
Time Frame: post-operative week 1, post-operative month 1, and post-operative month 3
Population: The SPSS software package (version 17.0, SPSS Inc, Chicago, IL, USA) was used for statistical analysis and sample size calculation. Mean ultrasound time (UST), surgical time, cumulative dissipated energy (CDE), total BSS volume, and SIA were compared using multifactor analysis of variance.
Measure: Mean (Standard Deviation); unit: % of endothelial cell loss
Arm/Group | Group I | Group II | Group III
Number analyzed (Participants) | 40 | 40 | 40
% of endothelial cell loss
  Post-op 1m | 11.78 (7.27) | 13.03 (8.33) | 12.05 (9.31)
  Post-op 1 w | 7.77 (3.76) | 9.35 (4.69) | 7.93 (3.67)
  Post-op 3 month | 17.83 (5.65) | 18.08 (7.93) | 17.66 (5.26)

2. Secondary Outcome: Best-corrected Visual Acuity
Description: The best-corrected visual acuity (BCVA) was measured, using an ETDRS chart and auto-refraction as refined by an ophthalmologist, preoperatively and at postoperative 1 day, 1 week, 1 month and 3 months.
Time Frame: post-operative week 1, post-operative month 1, and post-operative month 3
Population: The SPSS software package (version 17.0, SPSS Inc, Chicago, IL, USA) was used for statistical analysis.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Group I | Group II | Group III
Number analyzed (Participants) | 40 | 40 | 40
logMAR
  Pre-op 1 day | 0.16 (0.10) | 0.13 (0.11) | 0.15 (0.11)
  Post-op 1 day | 0.66 (0.27) | 0.71 (0.20) | 0.73 (0.23)
  Post-op 1 month | 0.89 (0.20) | 0.91 (0.13) | 0.88 (0.14)
  Post-op 3 months | 0.98 (0.11) | 1.01 (0.09) | 0.98 (0.10)

3. Primary Outcome: Surgically Induced Astigmatism
Description: Corneal astigmatism was measured using an eye scanner (Pentacam; Oculus, Wetzlar, Germany), and the SIA was calculated at each postoperative visit using the following equation.
Time Frame: post-operative week 1, post-operative month 1, and post-operative month 3
Measure: Mean (Standard Deviation); unit: Diopters
Arm/Group | Group I | Group II | Group III
Number analyzed (Participants) | 40 | 40 | 40
Diopters
  Post-op 1 day | 1.2 (0.32) | 0.91 (0.34) | 0.951 (0.28)
  Post-op 1 week | 0.61 (0.24) | 0.74 (0.25) | 0.79 (0.23)
  Post-op 1 month | 0.4 (0.21) | 0.46 (0.24) | 0.75 (0.31)
  Post-op 3 months | 0.26 (0.18) | 0.31 (0.19) | 0.66 (0.21)

ADVERSE EVENTS:
Description: Total Number of Participants at Risk for this Observational Study (e.g., serious and/or other [non-serious] adverse events were not collected/assessed).
Arm/Group | Group I | Group II | Group III
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less